CLINICAL TRIAL: NCT02642263
Title: Effect of the Uterotonic Carbetocin on Acute Post Cesarean-Section Pain, A Prospective Randomised Study
Brief Title: Effect of the Uterotonic Carbetocin on Acute Post Cesarean-Section Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uterotonic Carbetocin
Record Dates: First submitted 2015-12-21; First posted 2015-12-30 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Cesarean Delivery
MeSH Terms: interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (No Intervention): Oxytocin 20 IE in 500 ml G Na intravenous infusion over 6 hours (GlucoSalin 2:1; 2/3 glucose 5%+1/3 NaCl 0.9%), Sintetica-Bioren, Switzerland, after birth of the baby. For blinding purposes a 3ml NaCl 0.9% syringe is administered intravenously after birth of the baby as well.
- Carbetocin (Experimental): 100 mcg of Carbetocin, Ferring, Switzerland, as iv administration after birth of the baby. For blinding purposes an intravenous infusion of 500 ml G Na (GlucoSalin 2:1; 2/3 glucose 5%+1/3 NaCl 0.9%) is administered over 6 hours.
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — Postpartum uterotonic drug
  Other Names: Pabal, Ferring, Baar, Switzerland
  Arms: Carbetocin

SUMMARY:
Carbetocin is an oxytocin agonist used for prevention of postpartum bleeding after cesarean delivery. First studies revealed in 2012 an analgesic effect of carbetocin, compared to its parent substance oxytocin. This study will enroll 78 women undergoing cesarean delivery. In a double-blind, prospective design patients will be either attributed to the oxytocin or the carbetocin study arm. The primary endpoint will be the area of hyperalgesia around the cesarean delivery scar. This will be performed with a von Frey hair, resulting in a unpleasant feeling in the area of hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45, uneventful pregnancy, on term (>37 0/7 weeks of gestation), scheduled elective CS including repeat CS

Exclusion Criteria:

* lack of informed consent, active labor, multiple pregnancy, polyhydramnios, severe fetal malformations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Cesarean delivery scar cutaneous hyperalgesia | 4 hours after cesarean delivery
  In the area of the cesarean delivery scar, the area of dynamic secondary hyperalgesia for punctate mechanical stimuli around the surgical incision will be measured around her scar according to the method described by Stubhaug et al. In brief, stimulation with a Von Frey Filament (225.1gr) is started from outside the hyperalgesic area where no pain sensation is experienced toward the incision until the patient reports a distinct change in perception. The first point where a painful, sore, or sharp feeling appears is recorded, and the distance to the incision is measured. If no change in sensation appears, stimulation is stopped at 0.5 cm from the incision. The area of secondary hyperalgesia is determined by testing along radial lines separated by 5 cm around the incision. The observations are translated onto graph paper, and the surface is calculated as cm2/cm of incision.

SECONDARY OUTCOMES:
Pressure pain detection threshold | before cesarean
  Pain detection thresholds will be measured with an electronic pressure algometer (Algometer, Somedic, Denmark) applied at the center of the pulp of the 2nd toe. The probe has a surface area of 1 cm2. The pressure is increased from 0 at a rate of 30kPa/s to a maximum pressure of 1000kPa. Pain detection threshold is defined as the point at which the pressure sensation turns to pain. The subjects are instructed to press a button when these points are reached. The algometer displays the pressure intensity at which the button is pressed. If the subjects do not press the button at a pressure of 1000 kPa, this value is considered as threshold.
Pressure pain detection threshold | 4 hours after cesarean
  Pain detection thresholds will be measured with an electronic pressure algometer (Algometer, Somedic, Denmark) applied at the center of the pulp of the 2nd toe. The probe has a surface area of 1 cm2. The pressure is increased from 0 at a rate of 30kPa/s to a maximum pressure of 1000kPa. Pain detection threshold is defined as the point at which the pressure sensation turns to pain. The subjects are instructed to press a button when these points are reached. The algometer displays the pressure intensity at which the button is pressed. If the subjects do not press the button at a pressure of 1000 kPa, this value is considered as threshold.
Pressure pain detection threshold | 24 hours after cesarean
  Pain detection thresholds will be measured with an electronic pressure algometer (Algometer, Somedic, Denmark) applied at the center of the pulp of the 2nd toe. The probe has a surface area of 1 cm2. The pressure is increased from 0 at a rate of 30kPa/s to a maximum pressure of 1000kPa. Pain detection threshold is defined as the point at which the pressure sensation turns to pain. The subjects are instructed to press a button when these points are reached. The algometer displays the pressure intensity at which the button is pressed. If the subjects do not press the button at a pressure of 1000 kPa, this value is considered as threshold.
Pressure pain detection threshold | 48 hours after cesarean
  Pain detection thresholds will be measured with an electronic pressure algometer (Algometer, Somedic, Denmark) applied at the center of the pulp of the 2nd toe. The probe has a surface area of 1 cm2. The pressure is increased from 0 at a rate of 30kPa/s to a maximum pressure of 1000kPa. Pain detection threshold is defined as the point at which the pressure sensation turns to pain. The subjects are instructed to press a button when these points are reached. The algometer displays the pressure intensity at which the button is pressed. If the subjects do not press the button at a pressure of 1000 kPa, this value is considered as threshold.
Pressure pain detection threshold | 6 weeks after cesarean
  Pain detection thresholds will be measured with an electronic pressure algometer (Algometer, Somedic, Denmark) applied at the center of the pulp of the 2nd toe. The probe has a surface area of 1 cm2. The pressure is increased from 0 at a rate of 30kPa/s to a maximum pressure of 1000kPa. Pain detection threshold is defined as the point at which the pressure sensation turns to pain. The subjects are instructed to press a button when these points are reached. The algometer displays the pressure intensity at which the button is pressed. If the subjects do not press the button at a pressure of 1000 kPa, this value is considered as threshold.
Baseline depression detection | before cesarean
  Beck Depression Inventory (BDI-II): a 21 question multiple choice inventory used to measure severity of depression. This will be used in order to assess an eventual prepartum depression, this measure aims at eliminating bias if detecting a postpartum depression by the Edinburgh Depression questionnaire
Postpartum depression | 6 weeks post cesarean
  Assessment of postpartum depression with the Edinburgh Postnatal Depression Scale. It is a 10 item questionnaire.
Cesarean delivery scar cutaneous hyperalgesia | 24 hours after cesarean
  In the area of the cesarean delivery scar, the area of dynamic secondary hyperalgesia for punctate mechanical stimuli around the surgical incision will be measured around her scar according to the method described by Stubhaug et al. In brief, stimulation with a Von Frey Filament (225.1gr) is started from outside the hyperalgesic area where no pain sensation is experienced toward the incision until the patient reports a distinct change in perception. The first point where a painful, sore, or sharp feeling appears is recorded, and the distance to the incision is measured. If no change in sensation appears, stimulation is stopped at 0.5 cm from the incision. The area of secondary hyperalgesia is determined by testing along radial lines separated by 5 cm around the incision. The observations are translated onto graph paper, and the surface is calculated as cm2/cm of incision.
Cesarean delivery scar cutaneous hyperalgesia | 48 hours after cesarean
  In the area of the cesarean delivery scar, the area of dynamic secondary hyperalgesia for punctate mechanical stimuli around the surgical incision will be measured around her scar according to the method described by Stubhaug et al. In brief, stimulation with a Von Frey Filament (225.1gr) is started from outside the hyperalgesic area where no pain sensation is experienced toward the incision until the patient reports a distinct change in perception. The first point where a painful, sore, or sharp feeling appears is recorded, and the distance to the incision is measured. If no change in sensation appears, stimulation is stopped at 0.5 cm from the incision. The area of secondary hyperalgesia is determined by testing along radial lines separated by 5 cm around the incision. The observations are translated onto graph paper, and the surface is calculated as cm2/cm of incision.
Cesarean delivery scar cutaneous hyperalgesia | 6 weeks after cesarean
  In the area of the cesarean delivery scar, the area of dynamic secondary hyperalgesia for punctate mechanical stimuli around the surgical incision will be measured around her scar according to the method described by Stubhaug et al. In brief, stimulation with a Von Frey Filament (225.1gr) is started from outside the hyperalgesic area where no pain sensation is experienced toward the incision until the patient reports a distinct change in perception. The first point where a painful, sore, or sharp feeling appears is recorded, and the distance to the incision is measured. If no change in sensation appears, stimulation is stopped at 0.5 cm from the incision. The area of secondary hyperalgesia is determined by testing along radial lines separated by 5 cm around the incision. The observations are translated onto graph paper, and the surface is calculated as cm2/cm of incision.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Surbek, Prof, Study Director — Bern University Hospital
Locations (1):
- Dep. of Anesthesiology and Pain Medicine, Bern University Hospital, Bern, Switzerland